CLINICAL TRIAL: NCT05178667
Title: Effect of Carrot Seed and Rose Hip Extracts on Weight Management in Subjects With Overweight or Moderate Obesity. A Controlled, Randomized and Double-blind Study.
Brief Title: Food Supplement Effect on Overweight or Moderate Obesity
Acronym: PHYTOENIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Principal investigator, Institut Pasteur de Lille
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-A02422-39
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Contraceptives, Oral; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose (Experimental): 4 capsules with 1.6g of active product per day: 2 at breakfast and 2 at dinner
  Interventions: Dietary Supplement: High dose
- Low dose (Active Comparator): 4 capsules with 0.8g of active product per day: 2 at breakfast and 2 at dinner
  Interventions: Dietary Supplement: Low dose
- Maltodextrin (Placebo Comparator): 4 placebo capsules (maltodextrin) per day: 2 at breakfast and 2 at dinner
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: High dose — Food supplements are consumed during 3 months by healthy volunteers.
  Arms: High dose
Dietary Supplement: Low dose — Food supplements are consumed during 3 months by healthy volunteers.
  Arms: Low dose
Dietary Supplement: Maltodextrin — Food supplements are consumed during 3 months by healthy volunteers.
  Arms: Maltodextrin

SUMMARY:
The aim of this study is to assess the effect of a food supplement containing extracts of carrot and rose hip seeds on the weight of volunteers with overweight or moderate obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 kg / m² (limits excluded),
* Having a fat mass (measured by impedance balance in kg) according to the following table:

Men 18-29 years : ≥ 21.2 kg; Men 30-49 years : ≥ 21.6 kg; Men 50-65 years : ≥ 23.8 kg; Women 18-29 years : ≥ 31.4 kg; Women30-49 years : ≥ 31.8 kg; Women 50-65 years : ≥ 33.9 kg.

* Willing to observe dietetic plan in accordance with dietitian evaluation,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme.

Exclusion Criteria:

* Dyslipidemia or hyperlipidemia:

  * Fasting total cholesterol ≥ 3.0 g / L
  * Fasting triglycerides> 2.5 g / L
  * with heterozygous familial hypercholesterolemia,
* Diabetes treated or not with medication,
* With severe hepatic and / or renal impairment, liver enzyme level (ALT and / or AST) greater than 2.5 times the upper normal limit,
* TSH abnormal or not stable for at least 3 months,
* History of cardiac disease (heart attack, stroke, coronary artery disease) or chronic inflammatory disease in the previous 6 months,
* With cancer or having had cancer in the 3 years preceding the study, with the exception of basal cell cancers of the skin,
* Taking drugs known to have an impact on weight management (corticosteroids, neuroleptics, anti-HIV triple therapy, etc.) in the month preceding inclusion and / or likely to consume them during the test,
* Taking antibiotic therapy, anti-depressant treatment or treatment related to anxiety in the month preceding the study,
* Taking anti-depressant treatment or treatment related to anxiety Subject in a state of depression,
* Weight loss treatment in the previous 6 months or having followed a specific treatment promoting weight loss,
* Non stable weight during the last 6 months (>5% change in total weight),
* With metal implant (to allow DEXA measurement),
* Blood donation in the month before the start of the study and during the study,
* Consuming food supplements or functional foods known to have an influence on weight management in the month preceding the inclusion and / or likely to take during the test,
* Following or having followed a hypocaloric diet (energy intake <1,500 kCal / day) in the month preceding inclusion and / or likely to undertake this diet during the test,
* Following a particular diet (vegan),
* Diagnosed eating disorders (bulimia, anorexia nervosa, vomiting),
* Intense sport exercise practice (physical activity more than 4 hours per week) or not willing to maintain their exercise practises stable during the test,
* Smoking more than 5 cigarettes per day, unstable cigarettes consumption, or smoking cessation during 6 months preceding the inclusion or during the test,
* Bariatric surgery or who has a gastroplasty ring,
* Consuming more than 2 (women) or 3 (men) standard drinks of alcoholic beverage daily,
* Consuming illicit drugs,
* Using topical anti-cellulite treatments,
* For woman: Pregnant or planned to become, breastfeeding, with non-effective contraception,
* Known allergy to one of the component of the supplement (carrot and rose hip),
* Suffering from serious illnesses such as cancer, recent myocardial infarction, serious digestive pathologies or others diseases found to be inconsistent with the conduct of the study by the investigator,
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Any other condition which in the investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline weight at 3 months | 0 month (inclusion), 3 months
  Weight (unit: kg)

SECONDARY OUTCOMES:
Body mass composition by DEXA (dual energy x-ray absorptiometry) | 0 month (inclusion), 3 months
  Lean body mass, total fat mass, subcutaneous fat mass, visceral fat mass (unit: g)
Anthropometric parameters | 0 month (inclusion), 1 month, 2 months, 3 months
  Hip circumference, waist circumference and thigh circumference (unit: cm)
Fasting glycemia | 0 month (inclusion), 3 months
  Carbohydrate metabolism: Fasting glycemia (unit: g/l)
Insulinemia | 0 month (inclusion), 3 months
  Carbohydrate metabolism: Insulinemia (unit: mU/l)
HbA1c | 0 month (inclusion), 3 months
  Carbohydrate metabolism: HbA1c (unit: percent)
HOMA index | 0 month (inclusion), 3 months
  Carbohydrate metabolism: determination of the HOMA index (calculated)
Lipid metabolism | 0 month (inclusion), 3 months
  Total cholesterol, HDL, LDL, Triglycerides (unit: g/l)
Free fatty acids | 0 month (inclusion), 3 months
  Lipid metabolism: free fatty acids (unit: micromol/l)
Hepatic metabolism | 0 month (inclusion), 3 months
  Creatinine (unit: mg/l)
Transaminases | 0 month (inclusion), 3 months
  Hepatic metabolism: ASAT/ALAT (unit: UI/l)
Sedimentation rate | 0 month (inclusion), 3 months
  Blood parameters: Sedimentation rate (unit: mm)
Blood count | 0 month (inclusion), 3 months
  Blood parameters: Blood count (unit: G/L)
Thyroid Stimulating Hormone | 0 month (inclusion), 3 months
  TSH (Thyroid Stimulating Hormone) (unit: mUI/l)
High sensible C-reactive protein | 0 month (inclusion), 3 months
  CRPhs (high sensible C-reactive protein) (unit: mg/l)
Heart rate | 0 month (inclusion), 1 month, 2 months, 3 months
  Hemodynamic parameters: Heart rate (unit: Pul/min)
Blood pressure | 0 month (inclusion), 1 month, 2 months, 3 months
  Hemodynamic parameters: Systolic blood pressure (unit: mm Hg) and Diastolic blood pressure (unit: mm Hg)
Body mass composition by impedancemetry | 0 month (inclusion), 1 month, 2 months, 3 months
  Lean body mass and total fat mass (unit: percent)
Weight | 0 month (inclusion), 1 month, 2 months, 3 months
  Anthropometric parameters: weight (unit: kg)
Height | 0 month (inclusion), 1 month, 2 months, 3 months
  Anthropometric parameters: height (unit: cm)
Body Mass Index | 0 month (inclusion), 1 month, 2 months, 3 months
  Anthropometric parameters: determined Body Mass Index (unit: kg/m²)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lecerf, MD, Principal Investigator — Institut Pasteur de Lille - NutrInvest
Locations (2):
- France (2):
  - NutrInvest - Institut Pasteur de Lille, Lille, Nord
  - Institute of Cardiometabolism And Nutrition, Paris